CLINICAL TRIAL: NCT07230444
Title: Validation and Implementation With Artificial Intelligence of Software for the Intra-procedural Assessment of Uterine Artery EMBOlization
Brief Title: Artificial Intelligence for the Intra-procedural Assessment of Uterine Artery Embolization
Acronym: AI-EMBO
Status: Not yet recruiting | Type: Observational
Sponsor: Emanuele Barabino (Other)
Responsible Party: Sponsor-Investigator, Emanuele Barabino, Emanuele Barabino, MD, EBIR - Principal Investigator, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Organization: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Other Study IDs: AI-EMBO 2.0
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Uterine Fibroids (UF)
Keywords: uterine fibroids; embolization; uterine artery embolization; quantitative imaging; artificial intelligence
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 250 patients with a diagnosis of uterine fibroids who underwent uterine artery embolization: Women diagnosed with symptomatic uterine fibroids who underwent image-guided uterine artery embolization as treatment. No additional surgical or medical interventions were performed during the procedure.

SUMMARY:
Uterine artery embolization is a minimally invasive treatment for symptomatic uterine fibroids, but intra-procedural assessment of embolization adequacy currently relies on subjective angiographic criteria. This study evaluates a proprietary angiographic analysis software (AQ-VERO) that extracts quantitative time-to-density perfusion metrics in real time. The study aims to (1) validate the accuracy and reproducibility of AQ-VERO during uterine artery mebolization, and (2) develop an AI-based decision support system using AQ-VERO-derived metrics to improve objective intra-procedural assessment of treatment endpoints.

DETAILED DESCRIPTION:
Background and Rationale.

Uterine fibroids affect up to 70-80% of women of reproductive age. Uterine artery embolization achieves technical success rates above 95% and symptom improvement in approximately 75-90% of patients; however, it is associated with a 20-30% cumulative risk of clinical failure or need for reintervention at 5 years. Current intra-procedural assessment of embolization adequacy is based on qualitative angiographic criteria (e.g., "5-10 heartbeats stasis," "pruned tree appearance"), which are subjective and operator-dependent. Emerging evidence suggests that achieving near-complete, rather than complete, flow stasis may reduce post-procedural pain, underscoring the need for quantitative and standardized assessment tools.

AQ-VERO is an internally developed software platform that performs quantitative time-to-density (TTD) analysis of angiographic images to objectively quantify uterine and fibroid perfusion in real time.

Objectives.

Primary Objective: To validate the accuracy and intra-/interobserver reproducibility of AQ-VERO TTD metrics in quantifying perfusion changes during uterine artery embolization.

Secondary Objectives: (a) To develop and internally validate an AI-based decision support model that uses AQ-VERO-derived metrics to identify predefined embolization endpoints; (b) To explore the correlation between intra-procedural TTD metrics and post-procedural clinical outcomes, including symptom improvement, early pain scores, and need for reintervention.

Study Design. This is an ambispective (includes retrospective and prospective follow-up), multicenter observational study including women undergoing uterine artery embolization for symptomatic uterine fibroids. Standardized angiograms will be acquired and analyzed with AQ-VERO to extract TTD perfusion parameters (e.g., time-to-peak, area under the curve, wash-in/wash-out characteristics). Operators will document conventional qualitative angiographic endpoints. Clinical and imaging follow-up will be collected according to institutional protocols.

Primary Objective:

• To evaluate whether the AI predictive model developed using AQ-VERO© metrics can predict the clinical outcome, defined as complete or significant resolution of fibroid-related symptoms.

Secondary Objectives:

* To correlate distinct TTD curve morphologies and AQ-VERO metrics with post-procedural pain.
* To detect the presence of collateral or accessory arterial supply that may compromise embolization efficacy.

Significance. This study is expected to establish a quantitative and AI-augmented framework for intra-procedural embolization assessment during uterine artery embolization, potentially reducing variability and improving long-term clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥18 years
* Symptomatic uterine fibroids (e.g., bleeding, bulk symptoms, pain)
* Underwent UAE as definitive therapy
* Availability of baseline clinical/imaging data (for retrospective arm) or ability to provide informed consent (for prospective arm)

Exclusion Criteria:

* Lack of clinical follow-up
* Poor quality or incomplete angiographic images.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of adult female patients aged 18 to 55 years with symptomatic uterine fibroids who underwent or are undergoing uterine artery embolization as their primary treatment. All participants must have angiographic imaging suitable for quantitative analysis and a minimum of 6 months of available clinical follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the AUPRC of the predictive models. | From treatment to the end of the required follow-up (6 months).
  The Area Under the Precision-Recall Curve (AUPRC) will be calculated to evaluate the performance of the AI-based decision support model in identifying clinically relevant embolization endpoints. AUPRC is a threshold-independent metric that summarizes the tradeoff between precision (positive predictive value) and recall (sensitivity) across all decision thresholds. It is particularly suitable for imbalanced datasets, where positive outcome events may be less frequent. Higher AUPRC values indicate better discriminative performance of the model.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Cittadini, MD, Study Chair — IRCCS Ospedale Policlinico San Martino
Locations (1):
- IRCCS OSpedale Policlinico San Martino, Genova, Genova, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.

REFERENCES:
- [Result] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Result] Pron G, Bennett J, Common A, Wall J, Asch M, Sniderman K; Ontario Uterine Fibroid Embolization Collaboration Group. The Ontario Uterine Fibroid Embolization Trial. Part 2. Uterine fibroid reduction and symptom relief after uterine artery embolization for fibroids. Fertil Steril. 2003 Jan;79(1):120-7. doi: 10.1016/s0015-0282(02)04538-7. PMID 12524074
- [Result] Manyonda I, Belli AM, Lumsden MA, Moss J, McKinnon W, Middleton LJ, Cheed V, Wu O, Sirkeci F, Daniels JP, McPherson K; FEMME Collaborative Group. Uterine-Artery Embolization or Myomectomy for Uterine Fibroids. N Engl J Med. 2020 Jul 30;383(5):440-451. doi: 10.1056/NEJMoa1914735. PMID 32726530